CLINICAL TRIAL: NCT03920241
Title: Changes in Cognitive and Emotional Patterns Associated to Meditation and Compassion Training: Attentional Changes and Network Dynamics
Brief Title: Cognition and Emotion in Meditation: A Comparison Between Mindfulness and Compassion Standardized Programs
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carmelo Vázquez, Full Professor of Psychopathology, Universidad Complutense de Madrid
Other Study IDs: PSI-559959-R
Record Dates: First submitted 2019-03-12; First posted 2019-04-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Well-being; Emotion Regulation; Cognitive Control; Attention; Psychological Distress; Psychophysiologic Reaction; Compassion; Mindfulness
Keywords: Mindfulness; Compassion; Well-being; Network analysis; MBSR; CCT; Attentional blink; Cognition
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Stress Reduction; Control Groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MBSR group: Attendants to Mindfulness-Based Stres Reduction programs offered to the community by Complutense University
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- CCT group: Attendants to Compassion Cultivation Training programs offered to the community by Complutense University
  Interventions: Behavioral: Compassion Cultivation Training
- Control group: Control group matched by age, gender, and meditation experience.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The MBSR is an 8-week standardized program (Kabat-Zinn, 1990) consisted of 2.5-hour of face-to-face weekly sessions, and 45 minutes of daily home formal and informal practices. Training will be conducted in groups of 20-30 participants. During the program, different mindfulness practices are performed, including focused attention on the breath, open monitoring of awareness in body-scanning, prosocial meditation (i.e. loving kindness and compassion) and gentle yoga.
  Training is delivered by certificated instructors by the University of Massachusetts Centre for Mindfulness (https://www.umassmed.edu/cfm/).
  Other Names: MBSR
  Groups: MBSR group
Behavioral: Compassion Cultivation Training — The CCT is an 8-week standardized program (Jinpa, 2010; Jazaieri et al. 2013, 2014) consisting of 2.5-hour of face-to-face weekly sessions and 30 minutes of daily home formal and informal practices. Training will be conducted in groups of 20-30 participants. The CCT consists of six sequential steps: 1) Settling the mind and learn how to focus it; 2) Loving kindness and compassion for a loved one practice; 3) Loving kindness and compassion for oneself practice; 4) compassion toward others, embracing shared common humanity and developing appreciation of others; 5) compassion toward others including all beings; and 6) active compassion practices (Tonglen) which involve explicit evocation of the altruistic wish to do something about others' suffering.
  CCT program is delivered by certificated instructors by the University of Stanford Centre for Compassion and Altruism Research and Education (http://ccare.stanford.edu/).
  Other Names: CCT
  Groups: CCT group
Other: Control Group — A group of participants, matched by age, gender, and meditation experience is selected to compare their performance on experimental lab tasks in relation to the MBSR and CCT participants.
  Groups: Control group

SUMMARY:
The study is aimed at comparing the differential effects of two widely used standardized meditation programs: Mindfulness-Based Stress Reduction (MBSR) and Compassion Cultivation Training (CCT) in general population samples.

To address this goal, the effects will be measured by self-report questionnaires belonging to different domains (mindfulness, compassion, well-being, psychological distress, and psychological functioning) as well as information processing measures (i.e., Attentional Blink), and psychophysiological measures (EEG and EKG).

Changes will be assessed immediately after finishing the 8-week programs and through several inter-session assessments. Data analysis will include the mean change scores differences, as well as novel network analysis procedures to assess topological reorganization of constructs derived from the programs.

DETAILED DESCRIPTION:
The study has a twofold goal. Firstly, it will address whether the practice of different standardized meditation programs (MBSR and CCT) modify the distribution of limited attentional resources towards emotional information, measured by the performance in a variant of the Emotional Attentional Blink. Secondly, novel procedures of Network analysis will be used to examine whether the practice of different standardized meditation programs (mindfulness and compassion) impact on the network dynamics between mindfulness, compassion, well-being, psychological distress, and emotional and cognitive control constructs and how these constructs are eventually reorganized after the interventions.

There are two main corresponding hypotheses. First, meditation practice in general (both mindfulness and compassion) will change the attentional processing of emotional information, reflected by a significant reduction of the attentional blink deficit after the programs as compared to the performance of participants in matched Control group. Differences between both intervention groups will be analyzed. The second hypothesis states that, after meditation programs, the networks of these constructs will become topologically reorganized; more specifically, mindfulness, emotion regulation, and well-being constructs are expected to increase their centrality in the resulting network.

Procedure

The study will follow a pre-post design where participants will be blind to the aims of the study. Participants will be invited to participate at the moment they register in the official website offering the MBSR and CCT programs. After being recruited, those who accept to participate will fill out a brief online screening questionnaire on demographics and inclusion criteria and will sign an informed consent. Then participants will complete an online set of questionnaires (via Qualtrics software) of selected psychological domains associated to the main outcomes and variables studied in meditation literature (i.e., mindfulness, compassion, well-being, psychological distress, and emotional and cognitive control constructs). The online assessment will be completed the week before starting the program (baseline assessment) and during the week after the end of the MBSR (post-assessment). When necessary, reminders will be scheduled for those participants who have not completed the questionnaires. Each pre and post online evaluation will last approximately 45 minutes.

Participants are invited to attend a one-hour experimental session (i.e. Attentional Blink task) within the week before starting the meditation program. After completing a second informed consent, participants will fill out a set of questionnaires with mood (EEE), mindfulness (SM) and compassion (S_SC) state measure. Participants then will begin the Emotional Attentional Blink task divided into three blocks with a 1-minute break between the blocks. At the end of the task, participants will complete the "state measures" again and the session will end. After this lab session, participants will attend one of the two 8-week standardized meditation programs (MBSR or CCT). Finally, the same procedure will be followed for the post-experimental session within the week after the end of the programs. Each pre-post experimental session will last approximately one hour. After completing the post-treatment assessments, participants will be debriefed and will receive an individualized report of their questionnaires scores and the purposes of the study.

Programs description

The Mindfulness-Based Stress Reduction (MBSR) is an 8-week standardized program consisted of 2.5-hours of face-to-face weekly sessions, and 45 minutes of daily home formal and informal practices. Training will be conducted in groups of 20-30 participants. During the program, different mindfulness practices are performed, including focused attention on the breath, open monitoring of awareness in body-scanning, prosocial meditation (i.e. loving kindness and compassion) and gentle yoga.

The Compassion Cultivation Training (CCT) is also an 8-week standardized program consisting of 2.5-hours of face-to-face weekly sessions and 30 minutes of daily home formal and informal practices. Training will be conducted in groups of 20-30 participants. The CCT consists of six sequential steps: 1) Settling the mind and learn how to focus it; 2) Loving-kindness and compassion for a loved one practice; 3) Loving-kindness and compassion for oneself practice; 4) compassion toward others, embracing shared common humanity and developing appreciation of others; 5) compassion toward others including all beings; and 6) active compassion practices (Tonglen) which involve explicit evocation of the altruistic wish to do something about others' suffering. Finally, participants learn an integrative compassion practice combining the six essential elements into an integrative compassion meditation practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more
* Fluency in oral and written Spanish

Exclusion Criteria:

* Having any current of serious psychological disorder or substance abuse / dependence.
* Being currently enrolled in another standardized meditation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, from the community, attending courses of mindfulness or compasion at a University center.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in attention performance (Lab measures) | Pre- and post-intervention assessments (baseline and 8 weeks later)
  Attentional blink (accuracy emotion identification)
Change from Baseline in brain activity (Lab measures) | Pre- and post-intervention assessments (baseline and 8 weeks later)
  EEG (frontal lobe activity)
Change from Baseline in heart activity (Lab measures) | Pre- and post-intervention assessments (baseline and 8 weeks later)
  EKG (Heart rate variability)

SECONDARY OUTCOMES:
Mindfulness - General mindfulness | Pre and post-intervention assessments as well as intersession assessments (8 weekly assessments)
  Five-Facet Mindfulness Questionnaire (FFMQ)
Mindfulness - Non-attachment | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program))
  Non-Attachment Scale (NAS)
Mindfulness - Decentering | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Experiences Questionnaire (EQ)
Mindfulness - Interoceptive awareness | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Multidimensional assessment of interoceptive awareness (MAIA)
Mindfulness - State mindfulness | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  State Mindfulness Scale (SMS)
Compassion - Self-compassion | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Self-Compassion Scale (SCS)
Compassion - Compassion to others | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Compassion Scale (CS)
Compassion - Empathy | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Interpersonal Reactivity Index (IRI)
Compassion - State-compassion | Pre and post-intervention assessments as well as intersession assessments (weekly assessments during the 8 weeks of duration of the program)
  Self-Compassion Scale-State (SCS_S)
Psychological well-being - General well-being | Pre and post-intervention assessments (baseline and 8 weeks later)
  Pemberton Happiness Index (PHI)
Psychological well-being - Satisfaction with life | Pre and post-intervention assessments (baseline and 8 weeks later)
  Satisfaction With Life Scale (SWLS)
Psychological well-being - Optimism | Pre and post-intervention assessments (baseline and 8 weeks later)
  Life Orientation Test-Revised (LOT-R)
Psychological distress - feelings of depression, anxiety and stress | Pre and post-intervention assessments (baseline and 8 weeks later)
  Depression Anxiety Stress Scales (DASS-21)
Emotional and cognitive control - Rumination | Pre and post-intervention assessments (baseline and 8 weeks later)
  Ruminative Response Style (RRS)
Emotional and cognitive control - thought suppression | Pre and post-intervention assessments (baseline and 8 weeks later)
  White Bear Suppression Inventory (WBSI)
Emotional and cognitive control - Attentional control | Pre and post-intervention assessments (baseline and 8 weeks later)
  Attentional Control Scale (ACS)
Emotional and cognitive control - Emotion regulation | Pre and post-intervention assessments (baseline and 8 weeks later)
  Emotion Regulation Questionnaire (ERQ)
Emotional and cognitive control - Emotional States | Pre and post-intervention assessments (baseline and 8 weeks later)
  Emotional State Scale (ESS)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Vazquez, PhD, Principal Investigator — School of Psychology (Complutense University)
Locations (1):
- School of Psychology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Tang YY, Leve LD. A translational neuroscience perspective on mindfulness meditation as a prevention strategy. Transl Behav Med. 2016 Mar;6(1):63-72. doi: 10.1007/s13142-015-0360-x. PMID 27012254
- [Background] van der Velden AM, Roepstorff A. Neural mechanisms of mindfulness meditation: bridging clinical and neuroscience investigations. Nat Rev Neurosci. 2015 Jul;16(7):439. doi: 10.1038/nrn3916-c1. Epub 2015 Jun 17. No abstract available. PMID 26081785
- [Background] Kuyken W, Warren FC, Taylor RS, Whalley B, Crane C, Bondolfi G, Hayes R, Huijbers M, Ma H, Schweizer S, Segal Z, Speckens A, Teasdale JD, Van Heeringen K, Williams M, Byford S, Byng R, Dalgleish T. Efficacy of Mindfulness-Based Cognitive Therapy in Prevention of Depressive Relapse: An Individual Patient Data Meta-analysis From Randomized Trials. JAMA Psychiatry. 2016 Jun 1;73(6):565-74. doi: 10.1001/jamapsychiatry.2016.0076. PMID 27119968
- [Result] Malinowski P. Neural mechanisms of attentional control in mindfulness meditation. Front Neurosci. 2013 Feb 4;7:8. doi: 10.3389/fnins.2013.00008. eCollection 2013. PMID 23382709